CLINICAL TRIAL: NCT06434545
Title: SMEtH - Symptom Management Essentials at Home
Brief Title: Symptom Management Essentials at Home
Acronym: SMEtH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Zorgbelang Inclusief (Unknown); Comprehensive Cancer Centre The Netherlands (Other); ROC Midden Nederland (Unknown); University of Applied Sciences Utrecht (Other)
Responsible Party: Principal Investigator, Everlien de Graaf, Doctor, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 80-86300-98-060
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Symptom Management
Keywords: Symptom management; Palliative Care; Primary care; life-limiting illness; Palliative Reasoning

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group consists of 20 nursing team, each recruiting 20 clients with palliative care needs. This results in a total of 400 clients for the intervention group. A nursing team consists of nurse assistants, registered nurses and specialized nurses.
  Interventions: Behavioral: Palliative Reasoning methodology
- Control group (No Intervention): The control group consists of 20 nursing teams that will continue to provide care as previous to the start of the study. Contact persons also recruit 20 clients per nursing team, resulting in a total of 400 client for the control group.

INTERVENTIONS:
Behavioral: Palliative Reasoning methodology — Twenty nursing teams will be trained in the Palliative Reasoning methodology during a four hour training, split into two sessions. Additionally, teams receive a coaching session ones a month and practice with a real life case every week or two weeks during a one hour team meeting. This will be compared with 20 other nursing teams that will continue to provide care as usual.
  Arms: Intervention group

SUMMARY:
A cluster Randomized Controlled Trial (cRCT) that aims to determine the effect of the Palliative Reasoning (PR) methodology on the quality of life and symptom burden of patients dealing with a life-limiting illness and their loved ones, receiving palliative care services at home. Palliative Reasoning will be implemented from the first of may 2024 to 30 april 2025 in twenty nursing teams of a large homecare organization in Utrecht, the Netherlands, and will be compared with twenty control nursing teams. The effect of PR will be measured by means of questionnaires filled out by clients with a life expectancy of less than one year according to the surprise question "Would I be surprised if this person would die within one year?" and family caregivers. Parallel to the effect study, a process evaluation will be conducted in order to understand the implications of the results and its' societal and practical impact.

DETAILED DESCRIPTION:
The Palliative Reasoning (PR) methodology has been developed by University Medical Centre Utrecht (UMCU) in collaboration with the Netherlands Comprehensive Cancer organization (IKNL) to support nursing teams and other HCPs with the inter- and intradisciplinary communication and the early recognition, analysis and treatment of symptoms in patients requiring palliative care. This stepwise, iterative approach starts with HCPs identifying patients with palliative care needs by asking the surprise question "Would I be surprised if this patient would die within one year?". If the answer to the previous question is no, indicating not being surprised, a patient can be marked as being in a palliative phase of life. After the identification of the patient the method follows four steps: (1) Map out current symptoms, values, wishes and needs of patient and loved ones; (2) Analyze symptoms; (3) develop a proactive treatment plan; (4) Make agreements for the evaluation of the treatment plan.

After the training twenty of the forty nursing teams working for a large homecare organization, patients and family caregivers of both intervention teams and control teams can be included. The perceived symptom control, quality of life and symptom burden of patients and symptom burden of family caregivers, will be compared between intervention and control teams, to assess the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria client:

1. The client is 18 years or older.
2. The client is diagnosed with a life limiting illness or frailty syndrome with a life expectancy of less than a year, estimated by the nursing team, based on the Surprise Question.
3. The client lives at home and receives homecare
4. The client suffers from at least 1 symptom identified by means of the problem list of the Distress Thermometer.

Inclusion Criteria primary caregiver:

1. The primary caregiver is 18 years or older.
2. The primary caregiver has a relative with a life-limiting illness with a life expectancy <1 year.
3. Is able to speak and read Dutch

A nursing team is eligible when:

1. The nurses that are part of the nursing team are motivated to participate in the study.
2. The Nursing team consists of nurses that are sufficiently experienced in the work that they to effectively learn new competences during training sessions.

Exclusion Criteria:

Clients and primary caregivers that are diagnosed with cognitive impairment and/or unable to read and speak Dutch, will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Perceived symptom control of clients and family caregivers dealing with a life-limiting illness | One month after implementation
  This outcome will be measured by asking the participant "Do you feel your symptoms are under control?".

SECONDARY OUTCOMES:
Quality of life of clients dealing with a life-limiting illness | Assessed after one month, three months and six months after implementation.
  EORTC QLQ C15 will be used to determine the QoL.
Symptom burden of clients dealing with a life-limiting illness | Assessed at one month, three months and six months after implementation.
  Utrecht Symptom Diary Four Dimensional (USD4D) will be used to determine symptom burden. The USD4D comprises of questions regarding the physical, psychological, social, and spiritual dimension, which are rated on a scale from 0-10 (0 = symptom is absent to 10 = severity symptom is the worst imaginable).
Primary caregiver burden | Assessed at one, three and six months after implementation.
  The primary caregiver burden Is assessed by means of the Self Rated Burden Scale, which is a one item numerical scale answering the question "How do I perceive the care for my loved one at the moment?"(35-38). The question is answered on a scale of 0 to 10, in which 0 refers to "not at all straining" and 1 refers to "much to straining". In addition, the perceived burden of informal care (Dutch: Ervaren Druk Informele Zorg (EDIZ)) will be used, assessing aspects of informal care contributing to the perceived burden(39). The EDIZ is developed for the use in caregivers of patients suffering from dementia at home, however, this measurement instrument is widely used to assess the level of burden of caregivers of patients with a life-limiting illness. This instrument contains 9 statements to which patients must answer "no!", "no", "more or less", "yes" or "yes!".

OTHER OUTCOMES:
Client demographics | Questioned at baseline
  age, gender, marital status, education level, employment status (retired, unemployed, employed), (past) illness, type of employment (in the past), duration of illness, treatment, phase of illness, comorbidity, performance status (KPS), time under nursing care, number of visits per day/week.
Primary caregiver demographics | Questioned at baseline
  age, gender, education level, role, employment status assessed at enrollment.
Nursing team demographics | Questioned after baseline
  education level, local collaborations with GP and paramedics, symptom management practices.

CONTACTS AND LOCATIONS:
Overall Officials: Saskia Teunissen, Prof. dr., Study Director — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

DOCUMENTS (3):
  • Study Protocol (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT06434545/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT06434545/SAP_001.pdf
  • Statistical Analysis Plan (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT06434545/SAP_002.pdf